CLINICAL TRIAL: NCT02587767
Title: Prospective Randomized Controlled Clinical Trial to Evaluate the Effects of 577nm Micropulse Laser vs Half-dose Photodynamic Therapy on Acute Central Serous Chorioretinopathy
Brief Title: 577nm Micropulse Laser vs Half-dose Photodynamic Therapy on Acute Central Serous Chorioretinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Chen-jin, Dr, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 577MPLACS(Marshall Study)
Record Dates: First submitted 2015-10-17; First posted 2015-10-27 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Acute Central Serous Chorioretinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 577-MPL (Experimental): 577nm micropulse laser(577-MPL) will be performed of the areas identified on hyperfluorescent "hot spots" on the mid-phase (3 minutes) fluorescein.Multiple laser spots will be applied, covering the leakage area.
  Interventions: Device: 577-MPL
- HD-PDT (Active Comparator): Half-dose photodynamic therapy (HD-PDT) is administered to the patients. At 15 minutes after the start of the infusion, PDT laser treatment is performed with standard 50 J/cm2 fluency, a wavelength of 689nm, and a treatment duration of 83 seconds.
  Interventions: Device: HD-PDT

INTERVENTIONS:
Device: 577-MPL — All treatments were provided by a single practitioner with the 577-nm yellow laser system(Supra 577nm LaserSystem) in 577-MPL arm. The individual power for the patient was titrated at a normal area of near the affected area in micropulse model.The power titration was started at 700 milliwatt(mW) and then gradually increased until a just visible burn was seen. When this threshold was reached, the power was reduced by 50%, using a 100-μm spot diameter and a 200-ms duration with 5 % duty cycle.
  Arms: 577-MPL
Device: HD-PDT — 5 minutes after the start of the half-dose verteporfin infusion, the PDT treatment will been performed in HD-PDT arm. The treatment is performed with standard fluency (50 J/cm2), a PDT laser wavelength of 689 nm, and a standard treatment duration of 83 seconds.
  Arms: HD-PDT

SUMMARY:
The purpose of this study is to determine whether micropulse laser (MPL) is different to half-dose photodynamic therapy on acute central serous chorioretinopathy.

DETAILED DESCRIPTION:
Central serous chorioretinopathy(CSC) is characterized by serous detachment of neurosensory retina which can cause lose in visual acuity.Some studies have shown that Half-dose photodynamic therapy(PDT) is effective on CSC,although accompanied with side-effects,such as choroidal ischemia, retinal pigmental epithelium(RPE) atrophy,and RPE rip,and with exorbitant price.Recent retrospective studies suggest micropulse laser (MPL) therapy may also be effective without obvious complications in this disease. But to date, there is no study on effectiveness of CSC between PDT and MPL.

The study is the first prospective randomized controlled trial about 577nm micropulse laser versus half-dose photodynamic therapy on acute central serous chorioretinopathy.The null hypothesis of the study is that there is difference between MPL and half-dose photodynamic therapy on acute central serous chorioretinopathy at first month after treatment.The primary outcome measures is the proportion of eyes with complete absorption of subretinal fluid at 1 month after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. onset for the first time, as an episode duration of less than 6 months
2. patient was between 18 and 55 years of age
3. the presence of subretinal fluid(SRF) involving the macula and detected by use of optical coherence tomography (OCT)
4. active fluorescein leakage during fluorescein angiography (FA)
5. best corrected visual acuity (BCVA) more than 0.1, and less than 1.0

Exclusion Criteria:

1. previous PDT, focal photocoagulation, intravitreal injections of anti-vascular endothelial growth factor, or ocular surgery
2. other macular abnormalities such as choroidal neovascularization(CNV) or polypoidal choroidal vasculopathy(PCV)
3. retinal atrophy
4. pregnancy
5. inability to obtain photographs or to perform FA
6. use of steroid systemically or topically in the last 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
the proportion of eyes with complete absorption of subretinal fluid(SRF) | 1 month
  The primary outcome measure is the OCT-based improvement rate (defined as the proportion of eyes with complete absorption of subretinal fluid on OCT images

SECONDARY OUTCOMES:
Change of Best Corrected Visual Acuity(BCVA) | 1 month, 3 month, 6 month
Change of fundus autofluorescence | 1 month, 3 month, 6 month
  Fundus autofluorescence will be evaluated for different patterns（normal, increased, and decreased）before and after treatment
Change in 10°retinal sensitivity | 1 month, 3 month, 6 month
  Retinal sensitivity will be measured by microperimetry
the proportion of eyes with complete absorption of subretinal fluid(SRF) | 6 month
  The outcome measure is the OCT-based improvement rate (defined as the proportion of eyes with complete absorption of subretinal fluid on OCT images

CONTACTS AND LOCATIONS:
Overall Officials: Chenjin Jin, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University; Lijun Zhou, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
it is undecided to make individual participant data available when the study is going on